CLINICAL TRIAL: NCT00962507
Title: A Phase I Study Evaluating the Combination of the Deacetylase Inhibitor, LBH589 Plus the mTOR Inhibitor RAD001, in Relapsed and Refractory Adult Patients With Lymphoma
Brief Title: Panobinostat and Everolimus in Treating Patients With Relapsed or Refractory Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08099; P30CA033572 (NIH); CHNMC-08099 (Registry Identifier: PDQ); NOVARTIS-CHNMC-08099; CDR0000652208 (Registry Identifier: PDQ); NCI-2010-00259 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: recurrent adult T-cell leukemia/lymphoma; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; cutaneous B-cell non-Hodgkin lymphoma; Waldenstrom macroglobulinemia; refractory multiple myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Everolimus; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: everolimus — Beginning with 5 mg every other day Monday, Wednesday or Friday for a 28 day cycle. Dose escalation will be determined by the toxicities associated with treatment.
Drug: panobinostat — 10 mg every Monday and Thursday of a 28 day cycle. Dose escalation will be determined by the toxicities associated with treatment.
Other: laboratory biomarker analysis — Pre-study, day 1 and day 26 samples to evaluation how the study drugs work in vitro (in a test tube).
Other: pharmacological study — Pre-study, day 1 and day 26

SUMMARY:
RATIONALE: Panobinostat and everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Giving panobinostat together with everolimus may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of panobinostat when given together with everolimus in treating patients with relapsed or refractory lymphoma or multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and feasibility of combining panobinostat with everolimus in patients with recurrent or refractory lymphoma or multiple myeloma.
* To define the maximum tolerated dose of panobinostat in combination with everolimus in these patients.

Secondary

* To obtain preliminary data for response to this treatment regimen in these patients.
* To perform correlative studies relevant to this treatment regimen.

OUTLINE: This is a dose-escalation study of panobinostat.

Patients receive oral panobinostat 3 days a week and oral everolimus once every other day for 4 weeks Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples may be collected for pharmacokinetic and correlative laboratory studies.

After completion of study treatment, patients are followed up for ≥ 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Hodgkin or non-Hodgkin lymphoma (including small lymphocytic lymphoma [SLL])

    * Any histology, including B, T, or NK/T cell allowed
  * Multiple myeloma (MM)
* Relapsed or refractory disease

  * Patients with lymphoma must have relapsed after or be refractory to an upfront regimen (e.g., CHOP or ABVD) and a salvage regimen (e.g., ICE or ESHAP)

    * Patients with SLL should have relapsed after a fludarabine-containing regimen
  * Patients with MM must have progressed within 100 days after receiving a regimen containing bortezomib and either thalidomide or lenalidomide AND have a 25% increase in serum paraproteins, urinary light chains, or plasma cell number in the bone marrow
* No active CNS disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³ (transfusion allowed in patients with biopsy-proven bone marrow involvement)
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5.0 times ULN if elevation due to leukemic involvement)
* Serum bilirubin ≤ 1.5 times ULN
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Serum potassium normal
* Serum phosphorous normal
* Serum total calcium (corrected for serum albumin) or serum ionized calcium normal
* Serum magnesium normal
* TSH and free T4 normal (thyroid hormone replacement allowed)
* Fasting serum cholesterol ≤ 300 mg/dL (or ≤ 7.75 mmol/L) AND fasting triglycerides ≤ 2.5 times ULN (elevated levels allowed provided an appropriate lipid-lowering medication has been initiated)
* LVEF normal by MUGA or ECHO
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method (including barrier method) contraception during and for 3 months after completion of study treatment
* No impaired cardiac function, including any of the following:

  * QTc > 450 msec by screening ECG
  * Congenital long QT syndrome
  * History of sustained ventricular tachycardia
  * History of ventricular fibrillation or torsades de pointes
  * Bradycardia, defined as heart rate (HR) < 50 beats/min (pacemaker allowed provided HR ≥ 50 beats/min)
  * Myocardial infarction or unstable angina within the past 6 months
  * NYHA class III-IV congestive heart failure
  * Right bundle branch block and left anterior hemiblock (bifascicular block)
* No uncontrolled hypertension
* No unresolved diarrhea > CTCAE grade 1
* No impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral agents (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* No other concurrent severe or uncontrolled medical condition
* No other primary malignancy within the past 5 years other than curatively treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin
* No known HIV or hepatitis C positivity
* No significant history of non-compliance to medical regimens
* No known hypersensitivity to everolimus, other rapamycins (e.g., sirolimus or temsirolimus), or their excipients

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior autologous or allogeneic stem cell transplantation allowed
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy and recovered
* More than 1 week since prior and no concurrent immunization with live attenuated vaccines
* More than 4 weeks since prior valproic acid
* No other prior histone deacetylase inhibitors
* No concurrent chronic systemic corticosteroids or another immunosuppressive agent, other than for control of itching (as in cutaneous T-cell lymphoma)

  * Concurrent corticosteroids allowed provided patient has been on a stable dosage regimen for ≥ 2 weeks before study entry
  * Topical or inhaled corticosteroids allowed
* No concurrent drugs that may induce torsades de pointes
* No concurrent CYP3A4 inhibitors
* No concurrent radiotherapy or other anticancer therapy
* No concurrent grapefruit, grapefruit juice, or seville (sour) oranges
* No concurrent medications that may cause QTc prolongation
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 90 days post treatment start
Toxicity | 90 days post treatment start

SECONDARY OUTCOMES:
Pharmacokinetic and correlative studies | Day 1 and Day 26 of the first cycle of treament

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Popplewell, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California